CLINICAL TRIAL: NCT06511297
Title: Metabolic Control of Aging and Disease - the MetAGE Deep Phenotyping Cohort (Pro-Metage)
Brief Title: Metabolic Control of Aging and Disease - the MetAGE Deep Phenotyping Cohort
Acronym: Pro-Metage
Status: Recruiting | Type: Observational
Sponsor: Thomas Scherer (Other)
Collaborators: Medical University of Graz (Other); University of Graz (Other)
Responsible Party: Sponsor-Investigator, Thomas Scherer, Assoc. Prof. Dr. med., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1632/2024
Record Dates: First submitted 2024-07-09; First posted 2024-07-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Aging; Aging Problems; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, hair, saliva, mucosa cells, stool, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Lean, young adults
  Interventions: Diagnostic Test: comprehensive metabolic phenotyping
- Overweight, young adults
  Interventions: Diagnostic Test: comprehensive metabolic phenotyping
- Lean, older adults
  Interventions: Diagnostic Test: comprehensive metabolic phenotyping
- Overweight, older adults
  Interventions: Diagnostic Test: comprehensive metabolic phenotyping
- Nonagenerians Age ≥ 90: Note: Nonagenarian Group will only be phenotyped once
  Interventions: Diagnostic Test: comprehensive metabolic phenotyping

INTERVENTIONS:
Diagnostic Test: comprehensive metabolic phenotyping — The investigators will employ state of the art techniques to metabolically phenotype the study groups using brain, cardiac and whole body magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS), wearables, optical coherence tomography longitudinally. In addition, a battery of patient reported outcome measures will be used to explore psychosocial aspects of aging.

SUMMARY:
The goal of this prospective observational study is to identify and validate blood based aging biomarkers in relation to cardiometabolic phenotypes of young and old, female and male subjects with or without obesity.

The main question is to gain insights into the interaction of obesity related metabolic alteration and aging, and the relevance of loss of metabolic control in the development of age-related diseases in order to build a foundation for targeted drug- and lifestyle interventions in future studies.

DETAILED DESCRIPTION:
The ongoing increase in human life expectancy is steadily reshaping the demographic landscape, leading to a higher proportion of older adults, many of whom suffer from multiple health conditions. These unprecedented demographic shifts come at a significant socioeconomic cost, as aging stands as the primary risk factor for chronic disabilities and disorders such as cardiovascular diseases, dementia, type 2 diabetes, obesity, steatotic liver disease and infections. Consequently, promoting healthy aging emerges as one of the most pressing societal challenges in the foreseeable future, underscoring the urgent need for clinically validated strategies to extend the disease-free phase of life, known as health span.

The Pro-MetAGE prospective cohort as part of the clinical program of the MetAGE Cluster of Excellence (Austrian Science Fund # 10.55776/COE14) will focus on understanding the metabolic dysregulation associated with aging in a metabolic at-risk population. Metabolic control, which encompasses various aspects and is influenced by numerous aging indicators, might be the primary driver of age-related diseases. For instance, contemporary markers of biological age, such as epigenetic clocks based on DNA methylation and cellular senescence markers, correlate more closely with metabolic processes like nutrient sensing and mitochondrial function rather than genome stability or telomere length.

Aging entails a gradual deterioration of several fundamental metabolic processes, including lipostasis (fat metabolism), proteostasis (protein homeostasis), polyamine metabolism, and mitochondrial function. These intracellular changes are compounded by alterations in intercellular and interorgan communication, affecting brain-organ interactions and immune function. The decline in these crucial processes can disrupt the regulatory mechanisms of metabolic control in a manner influenced by sex and gender. Consequently, the loss of metabolic control may exacerbate other aging processes, setting off a detrimental cycle of accelerated aging.

Disruption in metabolic regulation caused by calorie-rich diets, disturbed circadian rhythms, or sedentary lifestyle can lead to a diverse set of health issues known collectively as metabolic syndrome. These medical conditions, including obesity, high blood pressure, elevated lipid levels, insulin resistance, and high blood sugar, contribute to the development of prevalent age-related diseases such as cardiovascular disease, type 2 diabetes, retinal degeneration and metabolic dysfunction-associated steatotic liver disease, formerly known as nonalcoholic fatty liver disease, affecting millions of older individuals globally. Additionally, there exists a significant link between metabolic imbalance and dysfunction in the immune system, resulting in heightened susceptibility to infections, diminished response to vaccinations, and various neuropsychiatric disorders, especially depression. Hence, understanding the mechanisms underlying metabolic dysregulation holds immense importance in devising preventive measures against some of the most debilitating age-related ailments.

The proposed research project aims to prospectively identify and validate aging biomarkers in relation to age- and sex-related cardiometabolic changes in young and old individuals, who are lean or obese/overweight (i.e. a metabolic at-risk population) with regard to lipostasis, proteostasis, polyamine metabolism, mitochondrial function, inflammation and cellular senescence. The goal is to gain insights into the interaction of obesity related metabolic alteration and aging, and the relevance of loss of metabolic control in the development of age-related diseases in order to build a foundation for targeted drug- and lifestyle interventions in future studies.

ELIGIBILITY:
Inclusion Criteria:

Group 1 - Lean, young adults (n = 150)

* Age 18 - 35 years
* Body mass index (BMI) ≥ 18.5 and ≤ 24.9 kg/m2 (≥ 12 months)

Group 2 - Overweight, young adults (n = 150)

* Age 18 - 35 years
* BMI ≥ 28kg/m2 (≥ 12 months)

Group 3 - Lean, older adults (n = 150)

* Age ≥ 60 years
* BMI ≥ 18.5 and ≤ 24.9 kg/m2 (≥ 3 years)

Group 4 - Overweight, older adults (n = 150)

* Age ≥ 60 years
* BMI ≥ 28 kg/m2 (≥ 3 years)
* Subgroup A (n=75): with pre-existent cardiovascular disease defined as: history of myocardial infarction or evidence of coronary artery disease irrespective of revascularization status or history of ischemic or hemorrhagic stroke or presence of peripheral artery disease or heart failure with preserved ejection fraction (NYHA Class I-II).
* Subgroup B (n=75): without pre-existent cardiovascular disease

Group 5 - Nonagenerians Age ≥ 90 (n = 50)

* Age ≥ 90 years
* BMI ≥ 18.5 kg/m2 (≥ 3 years)

Exclusion Criteria:

Group 1 - Lean, young adults (n = 150)

* Highly physical active (i.e. > 5 times sporting activity / week with moderate to high intensity [heart rate 140 - 200bpm])
* Special diets (i.e. ketogenic diet and time-restricted eating)
* Clinically significant metabolic or endocrine disorders
* Claustrophobia
* drug abuse, alcohol > 15 drinks/week
* Heart failure, cardiovascular disease, immunosuppressive therapies, chronic inflammatory diseases and active oncologic conditions
* Metal implants that prohibit 3T MRI
* Pregnancy or breastfeeding

Group 2 - Overweight, young adults (n = 150)

* Highly physical active (i.e. > 5 times sporting activity / week with moderate to high intensity [heart rate 140 - 200bpm])
* Special diets (i.e. ketogenic diet and time-restricted eating)
* Active anti-obesity treatment (e.g. glucagon-like peptide 1 (GLP-1) analogues, polyagonists, naltrexone and bupropion)
* Clinically significant metabolic or endocrine disorders
* Claustrophobia
* drug abuse, alcohol > 15 drinks/week
* Heart failure, cardiovascular disease, immunosuppressive therapies, chronic inflammatory diseases and active oncologic conditions
* Metal implants that prohibit 3T MRI
* Pregnancy or breastfeeding

Group 3 - Lean, older adults (n = 150)

* Highly physical active (i.e. > 5 times sporting activity / week with moderate to high intensity [heart rate 140 - 200bpm])
* Special diets (i.e. ketogenic diet and time-restricted eating)
* Diabetes, overt hypo/hyperthyroidism
* Claustrophobia
* drug abuse, alcohol > 15 drinks/week
* Metal implants that prohibit 3T MRI
* Known severe cardiovascular diseases (i.e. PAD IIa or higher, advanced heart failure = left ventricular ejection fraction (LVEF) < 35% or NYHA Class III-IV)
* No previous heart failure, cardiovascular disease, immunosuppressive therapies, chronic inflammatory diseases and active oncologic conditions up until the age of 35 years.
* Life-threatening conditions with a life expectancy of less than 1 year or any other condition that would jeopardize proband safety/adherence while participating in this trial.

Group 4 - Overweight, older adults (n = 150)

* Special diets (i.e. ketogenic diet and time-restricted eating)
* Diabetes, overt hypo/hyperthyroidism
* Active anti-obesity treatment (e.g. GLP-1 analogues, polyagonists, naltrexone and bupropion)
* Claustrophobia
* drug abuse, alcohol > 15 drinks/week
* Metal implants that prohibit 3T MRI
* No previous heart failure, cardiovascular disease, immunosuppressive therapies, chronic inflammatory diseases and active oncologic conditions up until the age of 35 years.
* Life-threatening conditions with a life expectancy of less than 1 year or any other condition that would jeopardize proband safety/adherence while participating in this trial.

Group 5 - "healthy" Nonagenerians Age ≥ 90 (n = 50)

* Claustrophobia
* Clinically significant cognitive impairment compromising study adherence
* Metal implants that prohibit 3T MRI
* Life-threatening conditions with a life expectancy of less than 1 year or any other condition that would jeopardize proband safety/adherence while participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample from eastern Austria.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Epigenetic clocks | every 3 years
  Epigenetic clocks be measured assessing DNA methylation in whole blood. The investigators speculate that the biological age is accelerated in obesity/overweight persons independent of chronological age.

SECONDARY OUTCOMES:
Magnetic resonance spectroscopy | every 3 years
  Hepatic lipid content
Magnetic resonance imaging | every 3 years
  Whole body fat distribution

OTHER OUTCOMES:
Vibration-controlled transient elastography | every 3 years
  Liver stiffness, Hepatic lipid content
Body composition | every 3 years
  Air Displacement Plethysmograph with BodPod
Continuous glucose monitoring | every 3 years
  Continuous blood glucose monitoring over 2 weeks will be performed
Retina scans | every 3 years
  Optical coherence tomography angiography
Physical activity | every 3 years
  Wrist-based actigraphy will be used to assess physical activity

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medical University of Graz, Graz, Styria
  - Medical University of Vienna, Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Undecided